CLINICAL TRIAL: NCT02407197
Title: International T1 Multicentre CMR Study
Brief Title: International T1 Multicentre CMR Outcome Study
Acronym: T1-CMR
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Eike Nagel, Global Chief Investigator, King's College London
Other Study IDs: 2011-T1-MC
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cardiomyopathy; Heart Failure; Coronary Artery Disease; Chronic Kidney Diseases; Inflammation; Fibrosis
Keywords: T1 mapping; CMR; Outcome; multicenter
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Coronary Artery Disease; Renal Insufficiency, Chronic; Inflammation; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myocardial fibrosis is the fundamental substrate for the development of heart failure.

Cardiovascular magnetic resonance (CMR) allows non-invasive assessment of myocardial fibrosis based on late gadolinium enhancement (LGE) and T1 mapping.

Patients: Prospective longitudinal observational multicenter study of consecutive patients with suspected or known non-ischemic cardiomyopathy.

Imaging: Non-invasive measures of myocardial fibrosis: native T1, extracellular volume fraction (ECV) and LGE.

Primary endpoints: all cause and cardiovascular mortality.

Secondary endpoints: arrhythmic composite and HF composite endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. adults > 18 years of age
2. clinical indication for CMR
3. able to provide informed consent

Exclusion criteria:

contraindications for cardiac magnetic resonance imaging due to MR unsafe devices or objects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult population with clinically indicated CMR study
Sampling Method: Probability Sample
Enrollment: 1629 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year
  number of deaths

SECONDARY OUTCOMES:
Rate of Arrhythmia | 1 year
  number of fatal or aborted sudden cardiac death events (including a documented appropriate shock from ICD)
Rate of HF events | 1 year
  Number of HF death and unplanned HF hospitalization
Rate of deaths due to cardiovascular causes | 1 year
  Number of composite of sudden cardiac death (SCD), death from HF, death from stroke or thromboembolic event

CONTACTS AND LOCATIONS:
Overall Officials: Eike Nagel, MD, PhD, Principal Investigator — King's College London
Locations (4):
- Vincent's University, Sydney, New South Wales, Australia
- German Heart Institute Berlin, Berlin, Germany
- United Kingdom (2):
  - Guy's and St. Thomas' Hospital Trust, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dabir D, Child N, Kalra A, Rogers T, Gebker R, Jabbour A, Plein S, Yu CY, Otton J, Kidambi A, McDiarmid A, Broadbent D, Higgins DM, Schnackenburg B, Foote L, Cummins C, Nagel E, Puntmann VO. Reference values for healthy human myocardium using a T1 mapping methodology: results from the International T1 Multicenter cardiovascular magnetic resonance study. J Cardiovasc Magn Reson. 2014 Oct 21;16(1):69. doi: 10.1186/s12968-014-0069-x. PMID 25384607
- [Result] Hinojar R, Foote L, Arroyo Ucar E, Jackson T, Jabbour A, Yu CY, McCrohon J, Higgins DM, Carr-White G, Mayr M, Nagel E, Puntmann VO. Native T1 in discrimination of acute and convalescent stages in patients with clinical diagnosis of myocarditis: a proposed diagnostic algorithm using CMR. JACC Cardiovasc Imaging. 2015 Jan;8(1):37-46. doi: 10.1016/j.jcmg.2014.07.016. Epub 2014 Dec 10. PMID 25499131
- [Result] Haslbauer JD, Lindner S, Valbuena-Lopez S, Zainal H, Zhou H, D'Angelo T, Pathan F, Arendt CA, Bug G, Serve H, Vogl TJ, Zeiher AM, Carr-White G, Nagel E, Puntmann VO. CMR imaging biosignature of cardiac involvement due to cancer-related treatment by T1 and T2 mapping. Int J Cardiol. 2019 Jan 15;275:179-186. doi: 10.1016/j.ijcard.2018.10.023. Epub 2018 Oct 11. PMID 30360992
- [Result] Puntmann VO, Carr-White G, Jabbour A, Yu CY, Gebker R, Kelle S, Rolf A, Zitzmann S, Peker E, D'Angelo T, Pathan F, Elen, Valbuena S, Hinojar R, Arendt C, Narula J, Herrmann E, Zeiher AM, Nagel E; International T1 Multicentre CMR Outcome Study. Native T1 and ECV of Noninfarcted Myocardium and Outcome in Patients With Coronary Artery Disease. J Am Coll Cardiol. 2018 Feb 20;71(7):766-778. doi: 10.1016/j.jacc.2017.12.020. PMID 29447739
- [Result] Child N, Suna G, Dabir D, Yap ML, Rogers T, Kathirgamanathan M, Arroyo-Ucar E, Hinojar R, Mahmoud I, Young C, Wendler O, Mayr M, Sandhu B, Morton G, Muhly-Reinholz M, Dimmeler S, Nagel E, Puntmann VO. Comparison of MOLLI, shMOLLLI, and SASHA in discrimination between health and disease and relationship with histologically derived collagen volume fraction. Eur Heart J Cardiovasc Imaging. 2018 Jul 1;19(7):768-776. doi: 10.1093/ehjci/jex309. PMID 29237044
- [Result] Puntmann VO, Isted A, Hinojar R, Foote L, Carr-White G, Nagel E. T1 and T2 Mapping in Recognition of Early Cardiac Involvement in Systemic Sarcoidosis. Radiology. 2017 Oct;285(1):63-72. doi: 10.1148/radiol.2017162732. Epub 2017 Apr 27. PMID 28448233
- [Result] Hinojar R, Foote L, Sangle S, Marber M, Mayr M, Carr-White G, D'Cruz D, Nagel E, Puntmann VO. Native T1 and T2 mapping by CMR in lupus myocarditis: Disease recognition and response to treatment. Int J Cardiol. 2016 Nov 1;222:717-726. doi: 10.1016/j.ijcard.2016.07.182. Epub 2016 Aug 3. PMID 27521546
- [Result] Puntmann VO, Carr-White G, Jabbour A, Yu CY, Gebker R, Kelle S, Hinojar R, Doltra A, Varma N, Child N, Rogers T, Suna G, Arroyo Ucar E, Goodman B, Khan S, Dabir D, Herrmann E, Zeiher AM, Nagel E; International T1 Multicentre CMR Outcome Study. T1-Mapping and Outcome in Nonischemic Cardiomyopathy: All-Cause Mortality and Heart Failure. JACC Cardiovasc Imaging. 2016 Jan;9(1):40-50. doi: 10.1016/j.jcmg.2015.12.001. PMID 26762873
- [Result] Hinojar R, Varma N, Child N, Goodman B, Jabbour A, Yu CY, Gebker R, Doltra A, Kelle S, Khan S, Rogers T, Arroyo Ucar E, Cummins C, Carr-White G, Nagel E, Puntmann VO. T1 Mapping in Discrimination of Hypertrophic Phenotypes: Hypertensive Heart Disease and Hypertrophic Cardiomyopathy: Findings From the International T1 Multicenter Cardiovascular Magnetic Resonance Study. Circ Cardiovasc Imaging. 2015 Dec;8(12):e003285. doi: 10.1161/CIRCIMAGING.115.003285. PMID 26659373
- [Result] Isted A, Grigoratos C, Bratis K, Carr-White G, Nagel E, Puntmann VO. Native T1 in deciphering the reversible myocardial inflammation in cardiac sarcoidosis with anti-inflammatory treatment. Int J Cardiol. 2016 Jan 15;203:459-62. doi: 10.1016/j.ijcard.2015.10.199. Epub 2015 Oct 29. No abstract available. PMID 26547739
- [Result] Varma N, Hinojar R, D'Cruz D, Arroyo Ucar E, Indermuehle A, Peel S, Greil G, Gaddum N, Chowienczyk P, Nagel E, Botnar RM, Puntmann VO. Coronary vessel wall contrast enhancement imaging as a potential direct marker of coronary involvement: integration of findings from CAD and SLE patients. JACC Cardiovasc Imaging. 2014 Aug;7(8):762-70. doi: 10.1016/j.jcmg.2014.03.012. Epub 2014 Jul 16. PMID 25051945
- [Result] Puntmann VO, Arroyo Ucar E, Hinojar Baydes R, Ngah NB, Kuo YS, Dabir D, Macmillan A, Cummins C, Higgins DM, Gaddum N, Chowienczyk P, Plein S, Carr-White G, Nagel E. Aortic stiffness and interstitial myocardial fibrosis by native T1 are independently associated with left ventricular remodeling in patients with dilated cardiomyopathy. Hypertension. 2014 Oct;64(4):762-8. doi: 10.1161/HYPERTENSIONAHA.114.03928. Epub 2014 Jul 14. PMID 25024285
- [Result] Rogers T, Dabir D, Mahmoud I, Voigt T, Schaeffter T, Nagel E, Puntmann VO. Standardization of T1 measurements with MOLLI in differentiation between health and disease--the ConSept study. J Cardiovasc Magn Reson. 2013 Sep 11;15(1):78. doi: 10.1186/1532-429X-15-78. PMID 24025486
- [Result] Puntmann VO, Voigt T, Chen Z, Mayr M, Karim R, Rhode K, Pastor A, Carr-White G, Razavi R, Schaeffter T, Nagel E. Native T1 mapping in differentiation of normal myocardium from diffuse disease in hypertrophic and dilated cardiomyopathy. JACC Cardiovasc Imaging. 2013 Apr;6(4):475-84. doi: 10.1016/j.jcmg.2012.08.019. Epub 2013 Mar 14. PMID 23498674
- [Result] Puntmann VO, D'Cruz D, Smith Z, Pastor A, Choong P, Voigt T, Carr-White G, Sangle S, Schaeffter T, Nagel E. Native myocardial T1 mapping by cardiovascular magnetic resonance imaging in subclinical cardiomyopathy in patients with systemic lupus erythematosus. Circ Cardiovasc Imaging. 2013 Mar 1;6(2):295-301. doi: 10.1161/CIRCIMAGING.112.000151. Epub 2013 Feb 12. PMID 23403334
- [Derived] Hoffmann J, Puntmann VO, Fiser K, Rasper T, Berkowitsch A, Carerj ML, Nagel E, Dimmeler S, Zeiher AM. Circulating Th17 and Th22 Cells Are Associated With CMR Imaging Biosignatures of Diffuse Myocardial Interstitial Remodeling in Chronic Coronary Artery Disease. Circ Res. 2020 Aug 14;127(5):699-701. doi: 10.1161/CIRCRESAHA.120.316619. Epub 2020 Jun 24. No abstract available. PMID 32576092
- [Derived] Winau L, Hinojar Baydes R, Braner A, Drott U, Burkhardt H, Sangle S, D'Cruz DP, Carr-White G, Marber M, Schnoes K, Arendt C, Klingel K, Vogl TJ, Zeiher AM, Nagel E, Puntmann VO. High-sensitive troponin is associated with subclinical imaging biosignature of inflammatory cardiovascular involvement in systemic lupus erythematosus. Ann Rheum Dis. 2018 Nov;77(11):1590-1598. doi: 10.1136/annrheumdis-2018-213661. Epub 2018 Aug 4. PMID 30077990
- See also: Related Info — https://www.cardiac-imaging.org/t1-outcome-study.html